CLINICAL TRIAL: NCT04052438
Title: Predictive Inmunological Study to Assess the Rate of Gestation, Abortion and Live Newborn in Patients With Recurrent Abortions and Recurrent Implantation Failure.
Brief Title: PREDICTIVE IMMUNOLOGICAL STUDY OF RECURRENT ABORTIONS AND IMPLANTATION FAILURE
Status: Completed | Type: Observational
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: 1405-MAD-026-JG
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Maternal-Fetal KIR-HLA-C Compatibility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with recurrent abortion.: More than three idiopathic involuntary miscarriages.
  Interventions: Diagnostic Test: HLA-C and KIR determination for patients, couples, oocyte or semen donors, abortive tissue and newborn.
- Patients with implantation failure.: More than three IVF abortions with good quality embryos or more than two abortions in oocyte donation cycles.
  Interventions: Diagnostic Test: HLA-C and KIR determination for patients, couples, oocyte or semen donors, abortive tissue and newborn.

INTERVENTIONS:
Diagnostic Test: HLA-C and KIR determination for patients, couples, oocyte or semen donors, abortive tissue and newborn.

SUMMARY:
The involvement of the immune system in the process of implantation and its modulation as a therapeutic line in these alterations, failure of implantation and repetition abortion are controversial and make it necessary to conduct clinical studies properly led and with a study population chosen by strict criteria in order to better understand the involvement of the different innate and adaptive immune mechanisms in the field of reproductive medicine and especially in clinically expressed failures recurrent implantation failure and recurrent abortions.

DETAILED DESCRIPTION:
A prospective pilot study is proposed in patients with recurrent implantation failure and recurrent abortions undergoing assisted reproductive techniques.

The main objective of this study is to determine the involvement of key effectors of innate immune response in the endometrium that induces a pro-inflammatory response, and to be able to know in particular what is the distribution of KIR receptors in the uNK and the HLA-C typing in patient-mother, egg/semen donors, male-father, abortive remains, live newborns.

To this end, the distribution of KIR and HLA-C receptors will be studied two arms/patient groups, divided from a population chosen according to inclusion/exclusion criteria:

* Group I: group recurrent abortions.
* Group II: group recurrent implementation failure. The study population will include subjects of older age (aged between 18 and 37 years) who will be divided into 2 total Study Arms N x 200 (n x 100 for each arm).

ELIGIBILITY:
Inclusion Criteria in recurrent implantation failure:

* Body mass index between 19 and 27 kg/m2
* Patients with 3 or more IVF failures following transfer of good quality embryos or with 2 or more failures following embryo transfer in egg donation cycles.
* At least one embryo transfer is required to have been made in a blastocyst state (embryo on day 5) and with the current partner/donor.
* Study of normal karitype..
* Normal thrombophilia study.
* Vaginal exudate (Chlamydia, ureaplasma) normal
* Normal immune study.
* No hormone treatment in the two months prior to inclusion in the study.

Inclusión criteria in recurrent abortion:

* Body mass index between 19 and 27 kg/m2
* Patients with 3 or more recurrent abortions, natural gestations or after transfer of good quality embryos (own or ovodonation)
* Study of normal karitype.
* Normal thrombophilia study.
* Vaginal exudate (Chlamydia, ureaplasma) normal
* Normal immune study.
* No hormone treatment in the two months prior to inclusion in the study.

Exclusion Criteria:

* Pregnant or lactating women.
* They cannot offer cooperation.
* Participation in a study or clinical trial during the 3 months prior to inclusion.
* Patients with fibromes.
* Patients with PCOS.
* Patients with some genetic alteration (altered karitype, cystic fibrosis, multiple sclerosis, rheumatoid arthritis...)
* Patients chronic infectious disease.
* Patients in maintenance treatment with immunosuppressants.
* Patients who have received systemic corticosteroids in the last 4 weeks.
* Patients diagnosed with chronic lymphoproliferative disease.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with a history of recurrent abortion or recurrent implantation failure
Study Population: Women with a history of recurrent abortion (more than 3 idiopathic involuntary abortions) or recurrent implantation failure (more than 3 failures of IVF cycles with good quality embryos or more 2 failures in cycles with donor eggs) that will undergo a cycle assisted reproduction
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Maternal genetic compatibility profile fetal KIR-HLA-C | 2 years
  KIR AA, KIR AB, KIR BB

CONTACTS AND LOCATIONS:
Overall Officials: Diana Alecsandru, Principal Investigator — IVI Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adams EJ, Parham P. Species-specific evolution of MHC class I genes in the higher primates. Immunol Rev. 2001 Oct;183:41-64. doi: 10.1034/j.1600-065x.2001.1830104.x. PMID 11782246
- [Result] Apps R, Murphy SP, Fernando R, Gardner L, Ahad T, Moffett A. Human leucocyte antigen (HLA) expression of primary trophoblast cells and placental cell lines, determined using single antigen beads to characterize allotype specificities of anti-HLA antibodies. Immunology. 2009 May;127(1):26-39. doi: 10.1111/j.1365-2567.2008.03019.x. PMID 19368562
- [Result] Arck PC, Hecher K. Fetomaternal immune cross-talk and its consequences for maternal and offspring's health. Nat Med. 2013 May;19(5):548-56. doi: 10.1038/nm.3160. Epub 2013 May 7. PMID 23652115
- [Derived] Alecsandru D, Barrio A, Garrido N, Aparicio P, Pellicer A, Moffett A, Garcia-Velasco JA. Parental human leukocyte antigen-C allotypes are predictive of live birth rate and risk of poor placentation in assisted reproductive treatment. Fertil Steril. 2020 Oct;114(4):809-817. doi: 10.1016/j.fertnstert.2020.05.008. Epub 2020 Jul 31. PMID 32741616